CLINICAL TRIAL: NCT02590861
Title: Improving Oral Health Function With Implant Supported Partial Dentures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal staffing issues
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510M78701
Record Dates: First submitted 2015-10-20; First posted 2015-10-29 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Partial Edentulism
Keywords: Partial Dentures; Dental Implants; Quality of Life; Partial Edentulism
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dental implant (Experimental): All participants will receive the same intervention, this is a single group study.
  Interventions: Procedure: Dental implant

INTERVENTIONS:
Procedure: Dental implant — All participants will receive the same intervention, this is a single group study.

SUMMARY:
Distal extension Partial Removable Dental Prostheses (PRDPs) are less stable than tooth supported PRDPs due to progressive resorption of the alveolar ridge, which alters the retention and support generated by alveolar bone height. In addition, long-term wearers suffer with progressive alveolar ridge resorption that contributes to greater instability. The loss of stability and retention under the PRDP can lead to difficulties during mastication and swallowing, because of movement of the partial denture. These difficulties force patients to self-select food substances that are softer and easier to chew and possibly create changes in social eating. Therefore, having a partial denture that is poorly retentive will impact their oral health related quality of life Oral Health Related Quality of Life (OHRQoL). The placement of a dental implant into the edentulous area will transform a conventional PRDP into an Implant Supported PRDP, which will improve the functional capacity of partial denture wearers, especially their ability to comminute harder food substances such as fruits and nuts. The purpose of this study is to quantitatively measure the functional differences of patients wearing conventional PRDP with patients wearing implant supported PRDPs and Oral Health Impact of patients wearing implant supported PRDPs. The hypothesis is that patient wearing implant supported PRDPs will have greater functional capacity than patients wearing conventional PRDPs.

DETAILED DESCRIPTION:
In the past few decades there has been predictions regarding the level of edentulism, and the need for prosthetic rehabilitation of the population. Although studies estimate a decline in the percentage of edentulism, and a decreased need for removable prostheses, this is predicted to be offset by a projected 79% increase in the population that is 55 years or older, the number of individuals with existing prostheses needing new prostheses and maintenance, and the professional and public health responsibility to serve this population regardless to the level of edentulism. In spite of these demographic predictions, the need for prosthodontics services, both fixed dental prostheses and removable dental prostheses will continue to an oral health concern, in part due to the an aging population that retains more of their teeth resulting in partial edentulism.

Prosthetic rehabilitation should not only replace missing teeth, but it should restore oral function and have a positive impact on Oral-Health-Related Quality of Life (OHRQoL) of our patients. As the population continues to age worldwide, and the U.S. specifically, it will become increasingly important to improve the OHRQoL for the segment of our population possessing removable prostheses with high stability, and highly retentive prosthetic services. Traditionally, both complete and partial removable dentures lack retention and stability, and one recommendation to improve the function has been to utilize dental implants to retain and stabilize the prosthesis. Although, several investigations have evaluated the OHRQoL patients wearing removable the preponderate emphasis of these studies has been on complete denture patients. In addition, OHRQoL studies are generated by patient self-reports, and limited evaluation of actual oral function has been compared to the patient self-reported function. This study will use the OHIP to evaluate the OHRQoL of patients with distal extension partial dentures, as well as, actually measure the patients chewing ability.

This prospective cohort study is designed to gather preliminary data on the improvement of patient satisfaction and oral function for individuals wearing distal extension partial dentures that are supported by smaller length dental implants. Thirty healthy male and female participants aged 18 to 65 will be treated at the University of Minnesota Dental School, in the Clinical Research Center. A lower partial denture will be fabricated using routine prosthodontic techniques. The participants will receive a 7 mm X 3.75 mm or a 8.5 mm X 4.1 mm tapered implant, A Locator Abutment will be used to connect the denture to the implant to improve the retention and stability of the partial denture. The chewing ability and chewing pattern will be evaluated with a jaw-tracking device and the masticatory muscle activity will be evaluated with surface Electromyography (EMG). OHRQoL, chewing function, and patient satisfaction will be measured at the 1, 2, 6, and 12-month recall appointments.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria
* posterior mandibular edentulism (on at least one side of the arch),
* age 18-65,
* general good health (self-reported),
* a minimum of six mandibular anterior teeth remaining,
* moderate to good periodontal health,
* speak and read English at a high school level,
* psychologically able to receive treatment.

Exclusion Criteria:

* The exclusion criteria
* smokers,
* poorly controlled diabetics,
* untreated caries,
* participants needing more than two crowns to support prosthesis,
* symptomatic TMD,
* cognitive impairment,
* diagnosis of psychiatric disorder,
* less than 25 mm interarch space,
* lingual tori,
* vertical bone height less than 10 mm,
* Class II and Class III maxillomandibular relationship,
* posterior bite collapse,
* loss of vertical dimension,
* Lekholm/Zarb grade C or more,
* Lekholm/Zarb grade 3 or more,
* the principle investigator decision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The number of participants with improved chewing function due to implant placement using Oral Health Impact Profile (OHIP) | 1-month, 2-month, 6-month, and 12-month
  The patient's chewing ability will be evaluated at 1-month, 2-month, 6-month, and 12-month recall appointments to evaluate patient satisfaction.The Oral Health Related Quality of life will be measured using the OHIP_14 instrument at the baseline, 1-month, 6-month, and 12-month recall appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Mays, DDS, MS, PhD, Principal Investigator — University of Minnesota

REFERENCES:
- [Background] Weintraub JA, Burt BA. Oral health status in the United States: tooth loss and edentulism. J Dent Educ. 1985 Jun;49(6):368-78. No abstract available. PMID 3891805
- [Background] Douglass CW, Shih A, Ostry L. Will there be a need for complete dentures in the United States in 2020? J Prosthet Dent. 2002 Jan;87(1):5-8. doi: 10.1067/mpr.2002.121203. PMID 11807476
- [Background] U.S. Bureau of the Census, Statistical Abstract of the United States: 1996. 116th ed. Washington, DC,; 1996. P15, Table II, No. 14.
- [Background] Cooper LF. The current and future treatment of edentulism. J Prosthodont. 2009 Feb;18(2):116-22. doi: 10.1111/j.1532-849X.2009.00441.x. PMID 19254301
- [Background] Douglass CW, Watson AJ. Future needs for fixed and removable partial dentures in the United States. J Prosthet Dent. 2002 Jan;87(1):9-14. doi: 10.1067/mpr.2002.121204. PMID 11807477
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Slade GD, Nuttall N, Sanders AE, Steele JG, Allen PF, Lahti S. Impacts of oral disorders in the United Kingdom and Australia. Br Dent J. 2005 Apr 23;198(8):489-93; discussion 483. doi: 10.1038/sj.bdj.4812252. PMID 15849587
- [Background] McKenna G, Allen F, Woods N, O'Mahony D, Cronin M, DaMata C, Normand C. Cost-effectiveness of tooth replacement strategies for partially dentate elderly: a randomized controlled clinical trial. Community Dent Oral Epidemiol. 2014 Aug;42(4):366-74. doi: 10.1111/cdoe.12085. Epub 2013 Nov 20. PMID 24251386
- [Background] Thomason JM, Kelly SA, Bendkowski A, Ellis JS. Two implant retained overdentures--a review of the literature supporting the McGill and York consensus statements. J Dent. 2012 Jan;40(1):22-34. doi: 10.1016/j.jdent.2011.08.017. Epub 2011 Sep 3. PMID 21911034
- [Background] Hamdan NM, Gray-Donald K, Awad MA, Johnson-Down L, Wollin S, Feine JS. Do implant overdentures improve dietary intake? A randomized clinical trial. J Dent Res. 2013 Dec;92(12 Suppl):146S-53S. doi: 10.1177/0022034513504948. Epub 2013 Oct 24. PMID 24158335
- [Background] Al-Imam H, Ozhayat EB, Benetti AR, Pedersen AM, Gotfredsen K. Oral health-related quality of life and complications after treatment with partial removable dental prosthesis. J Oral Rehabil. 2016 Jan;43(1):23-30. doi: 10.1111/joor.12338. Epub 2015 Aug 13. PMID 26268721
- [Background] Fueki K, Igarashi Y, Maeda Y, Baba K, Koyano K, Sasaki K, Akagawa Y, Kuboki T, Kasugai S, Garrett NR. Effect of prosthetic restoration on oral health-related quality of life in patients with shortened dental arches: a multicentre study. J Oral Rehabil. 2015 Sep;42(9):701-8. doi: 10.1111/joor.12297. Epub 2015 Mar 25. PMID 25818656
- [Background] Shaghaghian S, Taghva M, Abduo J, Bagheri R. Oral health-related quality of life of removable partial denture wearers and related factors. J Oral Rehabil. 2015 Jan;42(1):40-8. doi: 10.1111/joor.12221. Epub 2014 Aug 21. PMID 25146999
- [Background] Visscher CM, Lobbezoo F, Schuller AA. Dental status and oral health-related quality of life. A population-based study. J Oral Rehabil. 2014 Jun;41(6):416-22. doi: 10.1111/joor.12167. Epub 2014 Apr 4. PMID 24698541